CLINICAL TRIAL: NCT00621153
Title: Open-label, Randomised, 2-Arm Parallel Group, Multicentre, 8-week, Phase IV Study to Assess the Antihypertensive Efficacy and Safety of the Candesartan Cilexetil 16 mg and Hydrochlorothiazide 12.5 mg Combination Therapy in Comparison With Candesartan 16 mg Monotherapy in Hypertensive Adults
Brief Title: Candesartan Effect in Second Stage Arterial Hypertension
Acronym: CAESAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2452L00016
Record Dates: First submitted 2008-01-24; First posted 2008-02-22 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2009-04

CONDITIONS: Stage II Hypertension
Keywords: Candesartan Cilexetil; hydrochlorothiazide; severe hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Candesartan cilexetil 16mg monotherapy
  Interventions: Drug: Candesartan Cilexetil
- 2 (Experimental): Candesartan cilexetil 16mg/HCT combination therapy
  Interventions: Drug: Candesartan Cilexetil; Drug: Hydrochlorothiazide
- 3 (Active Comparator): candesartan cilexetil 32mg monotherapy
  Interventions: Drug: Candesartan Cilexetil
- 4 (Experimental): Candesartan Cilexetil 32 mg/HCT combination therapy
  Interventions: Drug: Hydrochlorothiazide; Drug: Candesartan Cilexetil

INTERVENTIONS:
Drug: Candesartan Cilexetil — Candesartan Cilexetil 16 mg oral
  Other Names: Atacand
  Arms: 1; 2
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 mg
  Other Names: HCTZ; Diazide
  Arms: 2; 4
Drug: Candesartan Cilexetil — Candesartan Cilexetil 32 mg oral
  Other Names: Atacand
  Arms: 3; 4

SUMMARY:
To compare the changes in mean sitting DBP from baseline after 4 weeks of therapy with either candesartan cilexetil/HCT combination therapy or candesartan cilexetil monotherapy regimen

ELIGIBILITY:
Inclusion Criteria:

* Stage II essential hypertension (SBP≥ 160 or DBP≥100 mmHg), untreated, or treated with a maximum of 2 class of antihypertensive drugs

Exclusion Criteria:

* Current serum-creatinine >3 mg/dL, Current serum-potassium >5.5 mmol/L, 16.
* Pregnant or lactating women or women of childbearing potential who were not protected from pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hoon Choi, Principal Investigator — Severance Hospital; Joonwoo Bahn, Study Director — AstraZeneca Korea
Locations (1):
- Research Site, Seoul, South Korea

REFERENCES:
- [Derived] Lee HY, Hong BK, Chung WJ, Lee BK, Lee SH, Jeon DW, Ahn YK, Kim D, Park CK, Kim SH, Jung HO, Kim BO, Choi D. Phase IV, 8-week, multicenter, randomized, active treatment-controlled, parallel group, efficacy, and tolerability study of high-dose candesartan cilexetil combined with hydrochlorothiazide in Korean adults with stage II hypertension. Clin Ther. 2011 Aug;33(8):1043-56. doi: 10.1016/j.clinthera.2011.07.002. Epub 2011 Aug 10. PMID 21831438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 253 enrolled, 20 screening failure, 223 randomised, 198 completed
Groups:
- Candesartan Cilexetil/Hydroclorozide Combination Therapy: candesartan cilexetil/Hydroclorozide combination therapy
- Candesartan Cilexetil Monotherapy: candesartan cilexetil monotherapy
Period: Overall Study
Arm/Group | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy
Started | 117 (randomised) | 116 (randomised)
Discontinued | 20 | 15
Completed | 97 (completed) | 101 (completed)
Not Completed | 20 | 15
Not completed — Safety Reason | 8 | 7
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy | Total
Number analyzed (Participants) | 117 | 116 | 233
Age Continuous [Mean (Standard Deviation); unit: years] | 51.00 (10) | 47.80 (10) | 48.90 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 75 | 78 | 153

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mean Sitting DBP From Baseline After 4 Weeks of Therapy
Description: Mean of the changed DBP from baseline after 4 weeks
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy
Number analyzed (Participants) | 111 | 113
mmHg | -17.0 (0.89) | -14.1 (0.88)

2. Secondary Outcome: Changes in Mean Sitting SBP From Baseline After 4 Weeks of Therapy
Description: Mean of the changed SBP from baseline after 4 weeks
Time Frame: 4 weeks
Reporting Status: Not Posted
Measure: Least Squares Mean; unit: mmHg

3. Secondary Outcome: Proportion of Patients Achieving Goal of Mean Trough Sitting DBP (<90 mmHg, But <80 mmHg for DM & Chronic Kidney Disease) and SBP (<140 mmHg, But <130 mmHg for DM & Chronic Kidney Disease) After 4 Weeks of Therapy
Description: Percent of the patients achieving goal DBP and SBP after 4 weeks
Time Frame: 4 weeks
Reporting Status: Not Posted
Measure: Number; unit: Participants

4. Secondary Outcome: Proportion of Patients Achieving Goal of Mean Trough Sitting DBP (<90 mmHg, But <80 mmHg for DM & Chronic Kidney Disease) and SBP (<140 mmHg, But <130 mmHg for DM & Chronic Kidney Disease) After 8 Weeks of Therapy
Description: Percent of patients achieving goal of DBP
Time Frame: 8 weeks
Reporting Status: Not Posted
Measure: Number; unit: Participants

5. Secondary Outcome: Changes in Mean Sitting SBP From Baseline After 8 Weeks of Therapy
Description: Changed SBP from baseline after 8 weeks
Time Frame: 8 weeks
Reporting Status: Not Posted
Measure: Least Squares Mean; unit: mmHg

6. Secondary Outcome: Changes in Hs-CRP Level From Baseline After 8 Weeks of Therapy
Description: Change of hs-CRP from basline after 8 weeks
Time Frame: 8 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mg/dl

7. Secondary Outcome: Occurrence of Adverse Events (AE) and Discontinuation of Study Medication Due to AE's From Baseline (Randomisation) to the End of the Study (8 Weeks)
Description: Occurred number of AE and disconinuation of study medication due to the AE from basline after 8 weeks
Time Frame: 8 weeks
Reporting Status: Not Posted
Measure: Number; unit: Participants

8. Secondary Outcome: Compliance Levels at 4 Weeks and 8 Weeks of Therapy
Description: Percent of the number of returened pills to the number of prescrited pills
Time Frame: 8 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: percent

ADVERSE EVENTS:
Arm/Group | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 6 | 3
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy
Breast clacifications (Renal and urinary disorders) | 0/111 | 1/113
Scrub typhus (Skin and subcutaneous tissue disorders) | 0/111 | 1/113
Anal fistula (Gastrointestinal disorders) | 1/111 | 0/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Candesartan Cilexetil/Hydroclorozide Combination Therapy | Candesartan Cilexetil Monotherapy
Dizziness (Nervous system disorders) | 6/111 | 3/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less